CLINICAL TRIAL: NCT05854238
Title: A Multicenter, Open, Single Design, Researcher-led, Phase 1 Exploratory Study to Evaluate the Safety and Efficacy of Vein of Marshall RF Ablation Using TIRA(VA510 and Other 3 Types) in Patients With Persistent Atrial Fibrillation
Brief Title: The Study for Evaluate of Safety and Efficacy of Vein of Marshall RF Ablation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated without extension as the approved period expired before enrollment completion. Few eligible subjects were found, and investigators agreed not to extend the study.
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Min Soo Cho, associate professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TIRA-VoM
Record Dates: First submitted 2023-04-21; First posted 2023-05-11 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Marshall vein ablation; radiofrequency catheter ablation; vein of Marshall ablation; VoM; TauPnu
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: multicenter, open, single design, researcher-led, exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TIRA-VoM (Experimental): treated with transcatheter RF ablation system (TIRA catheter with its supplemental devices)
  Interventions: Device: TIRA-VoM

INTERVENTIONS:
Device: TIRA-VoM — treat persistent atrial fibrillation
  * The ablation temperature range is 50-60℃
  * About 2 minutes per ablation
  Other Names: VA510, VA515, VA410, VA415; VoM

SUMMARY:
The goal of this clinical trial is to evaluate the initial safety and effectiveness of an investigational medical device.

Electrode catheter ablation of the Marshall vein is performed using TIRA, a clinical trial medical device for patients with persistent atrial fibrillation,

DETAILED DESCRIPTION:
By analyzing the collected data, the initial safety and efficacy of the electrode catheter ablation effect of the clinical trial medical device is evaluated. After the clinical trial, the initial safety and efficacy of the electrode catheter ablation are evaluated by analyzing the changes in electrical signals before and after the procedure and by monitoring patients.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria will be included.

* Men and women who are at least 20 years of age (80 years of age or older for geriatric patients).
* Patients requiring electrode ablation because of persistent arrhythmia despite use of antiarrhythmic drugs for more than 6 weeks
* Patients diagnosed with persistent atrial fibrillation after 2 consecutive electrocardiograms or 24-hour Holter test performed at least 1 week apart.
* Patients who have been on anticoagulants for more than 6 weeks or have taken equivalent safety measures.
* Patients with no evidence of intracardiac thrombus on transesophageal echocardiography, intracardiac echocardiography, or equivalent cardiac imaging (Cardiac CT) performed within 48 hours.
* Patients who have made a voluntary decision to participate in this study and have given written informed consent.
* Patients who are able to understand, follow instructions and participate for the full duration of the study.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded.

* Patients whose computed tomography (CT) or antecedent venography performed at the screening visit demonstrates no identifiable Marshall's vein.
* Patients who have undergone catheter ablation for atrial fibrillation within 6 months prior to the screening visit, or who have undergone a surgical Maze procedure at any time.
* Patients with a diagnosis of acute coronary syndrome within 3 months or who have undergone a stenting procedure or coronary artery bypass grafting in a coronary artery proximal to the anticipated procedure route at the time of the study.
* Patients with severe heart failure and those suffering from cardiogenic shock
* Those who are with less than 40% emissions Those with less than 40% of the ejection fraction
* Patients with hypertrophic cardiomyopathy
* Patients who have contraindications to contrast medias or anticoagulants
* Patients with evidence of intra-atrial thrombus on imaging studies performed within 1 month of the procedure Patients with evidence of blood clots in the atrium on imaging tests performed within 1 month of the procedure.
* Patients who have intracardiac malignant tumors and a life expectancy of 12 months or less
* Subjects with severe renal dysfunction (creatinine cleararnce < 30ml/min)
* Pregnant women, nursing mothers, and women who are planning to become pregnant or who may become pregnant during the study but are not using medically acceptable contraception
* Participation in other clinical trials within 30 days prior to screening Patients who participated in other clinical trials within 30 days prior to screening.
* In addition to the above, those who have clinical findings that the principal investigator or person in charge deems inappropriate for this study based on medical judgment. In addition to the above, those who have clinically signifcant findings that are considered inappropriate for this study as determined medically by the principal investigator or person in charge.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Changes of electrical signals around the Marshall vein(1) | Immediately after the procedure
  Pacing progress through unipolar electrogram between radiofrequency catheter and ground patch:
  Failure to conduction is evaluated as successful ablation.
Changes of electrical signals around the Marshall vein(2) | Immediately after the procedure
  Pacing progress through unipolar electrogram between radiofrequency catheter and ground patch:
  Failure to conduction is evaluated as successful ablation.
Changes of electrical signals around the Marshall vein | Immediately after the procedure
  Observation of changes in unipolar electrogram between radiofrequency catheter and ground patch before and after resection:
  The size of the unipolar electrogram voltage before and after the procedure is compared, and if the reduction is more than 80%, it is evaluated as a successful ablation.
Rate of adverse events as a measure of safety | Immediately after the procedure
  Rate of composite endpoint of MACE death, myocardial infarction, cardiac tamponade, device related acrdiac surgery, stroke

SECONDARY OUTCOMES:
Efficacy of procedures(1) | 1 month post-procedure
  The Standard 12 Lead ECG : Whether normal sinus rhythm is maintained after surgery
Efficacy of procedures(2) | 1 month post-procedure
  24-hour Holter monitoring : Recurrence rate of atrial tachycardia/atrial fibrillation more than 30 seconds after the procedure
Adverse event(safety of procedures)(1) | 1 month post-procedure
  All adverse event rate, including Serious Adverse Events (SAEs) and Serious Device Adverse Events (SADEs).
  : Myocardial infarction due to coronary artery damage, intracardiac conduction disorder, pericardial tamponade, cardiac surgery related to medical devices, stroke, death, etc.
Adverse event(safety of procedures)(2) | 1 month post-procedure
  CT : Whether there is contracture or narrowing of the pulmonary veins at the treatment site.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Soo Cho, MD, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Asan Medical Center, Seoul, Songpa-gu

IPD SHARING:
Plan to Share IPD: No